CLINICAL TRIAL: NCT07392931
Title: Safety and Efficacy of Racecadotril in the Treatment of Acute Watery Diarrhea in Children: A Randomized Controlled Trial
Brief Title: Safety and Efficacy of Racecadotril in Children With Acute Watery Diarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Punjab Rangers Teaching Hospital Lahore (Other)
Responsible Party: Principal Investigator, Own Abbas, Own Abbas, Punjab Rangers Teaching Hospital Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT-2026-01
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Acute Watery Diarrhea
Keywords: Racecadotril; Pediatric Diarrhea; Acute Gastroenteritis; Oral Rehydration Therapy; Children
MeSH Terms: interventions — racecadotril

STUDY DESIGN:
Intervention Model Description: A randomized, parallel-group, placebo-controlled clinical trial comparing racecadotril plus standard therapy with placebo plus standard therapy in children with acute watery diarrhea
Who Masked: Participant
Masking Description: This was a single-blind study in which participants were unaware of treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Racecadotril plus Standard Therapy (Experimental): Participants received racecadotril in addition to standard therapy, including oral rehydration therapy and intravenous fluids when clinically indicated.
  Interventions: Drug: Racecadotril
- Placebo plus Standard Therapy (Placebo Comparator): Participants received placebo along with standard therapy, including oral rehydration therapy and intravenous fluids when clinically indicated.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Racecadotril — Racecadotril was administered orally at a dose of 1.5 mg/kg three times daily as an adjunct to standard therapy for acute watery diarrhea.
  Arms: Racecadotril plus Standard Therapy
Other: Placebo — Placebo was administered orally along with standard therapy for acute watery diarrhea.
  Arms: Placebo plus Standard Therapy

SUMMARY:
Acute watery diarrhea is a common cause of illness and hospitalization in children under five years of age, particularly in developing countries. The mainstay of treatment is oral rehydration therapy, which prevents dehydration but does not reduce stool frequency or duration of diarrhea. Persistent diarrhea often leads to repeated hospital visits and increased healthcare burden.

This randomized controlled trial was conducted to evaluate the safety and efficacy of racecadotril as an adjunct to standard oral rehydration therapy in children aged 3 months to 5 years hospitalized with acute watery diarrhea. Participants were randomly assigned to receive either racecadotril in addition to standard therapy or placebo with standard therapy.

The primary outcomes assessed were reduction in stool frequency and improvement in stool consistency, along with duration of hospital stay. The study aimed to determine whether racecadotril provides additional clinical benefit when used alongside standard treatment in pediatric acute watery diarrhe

DETAILED DESCRIPTION:
Acute watery diarrhea is a leading cause of morbidity and hospitalization among children under five years of age. Although oral rehydration therapy (ORT) remains the cornerstone of management, it does not reduce stool output, frequency, or duration of diarrhea. Racecadotril is an antisecretory agent that reduces intestinal fluid secretion without affecting gastrointestinal motility and has been shown to be safe in pediatric populations.

This study was a single-center, randomized, placebo-controlled clinical trial conducted in the Pediatric Department of Punjab Rangers Teaching Hospital, Lahore. Children aged 3 months to 5 years of either gender presenting with acute watery diarrhea were enrolled after obtaining informed consent from parents or guardians. Acute diarrhea was defined as the passage of three or more watery stools within 24 hours with a duration of less than 72 hours.

Participants were randomized using a lottery method into two groups. The intervention group received racecadotril at a dose of 1.5 mg/kg three times daily as an adjunct to standard oral rehydration therapy and intravenous fluids when indicated. The control group received placebo along with the same standard therapy. The study was conducted under single-blind conditions.

Children with severe dehydration, chronic diarrhea, blood or mucus in stools, age below 3 months, or significant comorbidities were excluded. Clinical outcomes were assessed by monitoring stool frequency, stool consistency, and duration of hospital stay.

The study was conducted over a six-month period from June 2025 to November 2025. Ethical approval was obtained from the Ethical Committee of Punjab Rangers Teaching Hospital, Lahore. Data were analyzed using SPSS software, with results expressed as means, standard deviations, frequencies, and percentages.

ELIGIBILITY:
Inclusion Criteria:Children aged 3 months to 5 years Diagnosis of acute watery diarrhea Duration of illness ≤ 72 hours Written informed consent obtained from parents or legal guardians

Exclusion Criteria:Chronic diarrhea Severe malnutrition Severe dehydration requiring intensive care Known hypersensitivity to racecadotril Presence of serious underlying systemic illness Patient with bloody mucus containing diarrhea

-

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea | Up to 72 hours after initiation of treatment
  Time from initiation of treatment until passage of the last unformed stool.
Reduction in stool frequency | Within 12 hours of treatment initiation
  Change in the number of watery stools per day after initiation of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Own Abbas, Principal Investigator — Punjab Rangers Teaching Hospital Lahore
Locations (1):
- Punjab Rangers Teaching Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and confidentiality considerations.